CLINICAL TRIAL: NCT00993759
Title: Phae 2 Efficacy Trial of AV Lotion for the Prevention of Cold Illness in Human Subjects
Brief Title: Efficacy Study of A Lotion to Prevent Common Colds
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Dial Corporation (Industry)
Collaborators: Hill Top Research (Industry)
Responsible Party: Leslie Lockhart, PhD / Principal Scientist, The Dial Corporation, A Henkel Company
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TM&R-0108-09-TXC
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Common Cold; Healthy
Keywords: common cold; rhinovirus; prevention
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No treatment (No Intervention)
- 3804-250A lotion (Experimental)
  Interventions: Drug: 3804-250A

INTERVENTIONS:
Drug: 3804-250A — 3.2 ml applied topically after hand washing and at least every 3 hours while awake.
  Arms: 3804-250A lotion

SUMMARY:
The purpose of this of this study is to determine if 3804-250A can prevent the common cold caused by the rhinovirus when applied to the hands. The study will also evaluate whether 3804-250A can prevent rhinovirus infection or common cold illnesses.

The study will also evaluate the safety of 3804-250A.

DETAILED DESCRIPTION:
Rhinovirus infections are the most frequent cause of up to 80% of cold illness during the fall rhinovirus season. While viral upper respiratory tract infections are generally mild and self-limiting, they are associated with an enormous economic burden, both in lost productivity and in expenditures for treatment. Rhinovirus infection is frequently associated with medical complications that have substantial morbidity such as acute otitis media and exacerbation of asthma.

Marketed treatment options for common colds consist primarily of symptomatic cold remedies that have only most effects on specific cold symptoms. 3804-250A is a topical treatment under investigation for the prevention of rhinovirus-associated colds by interruption of person-to-person transmission.

The study is a randomized trial conducted during a 9-week period during the fall rhinovirus epidemic season. Healthy, normal subjects will be randomly assigned to one of two treatment groups:

1. AV Lotion or
2. No Treatment control.

Subjects in the 3804-250A group will use the treatment on a defined schedule. The No Treatment control group will maintain their regular hand washing routine.

All subjects will record the presence of cold illness symptoms daily. Subjects will return to the study site weekly during the study for specimen collection for rhinovirus PCR, evaluation of irritation, review and clarification of study diary entries, for review and assessment of compliance, collection of adverse events and replenishment of study supplies. In addition, for the first five weeks of the study, subjects in the AV Lotion group will attend a second weekly compliance visits in which diaries and test product consumption will be assessed for compliance and collection of adverse events. Photographs of the hands will be taken for subjects who are withdrawn for skin irritation. The incidence of cold illness, rhinovirus-associated cold illness and rhinovirus infection will be compared between the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Read and sign a copy of the approved Consent Form;
* 18-40 years of age;
* If a woman of child bearing potential (WOCBP) must have a negative urine pregnancy test and be using an effective method of birth control such as, but not limited to, birth control pills, contraceptive foam, diaphragm, IUD, vasectomized partner, abstinence, or condoms;
* Capable of compliance with the required study and sick visits (i.e., no planned travel commitments);
* Willing to follow study restrictions;
* Generally in good health based on medical history interview.

Exclusion Criteria:

* Current participation on any study;
* Participation in an investigational drug study within 30 days of enrollment;
* Participation within 30 days of enrollment on any study where the hands were the test site;
* Pregnancy (as determined by an urine pregnancy test), lactation or planning a pregnancy during the course of the study;
* Daily smoker;
* Current or significant history of sinusitis;
* Skin conditions on the hands or wrists that would interfere with the evaluations, such as scars, tattoos, uneven skin tones, or other conditions;
* Allergy to soaps, detergents, preservatives, citric acid, malic acid or ethanol;
* Immunological disorders (i.e., AIDS, HIV, systemic lupus erythematosis, rheumatoid arthritis);
* Current use or use within 7 days prior to randomization of any antibacterial medications for treatment of respiratory infections;
* Current use or use within 7 days enrollment of topical drugs (e.g. hydrocortisone or other corticosteroids) to treat skin conditions on the hands or wrists, except for localized treatment of minor cuts or scrapes;
* Occupational or other requirement for unusually frequent hand washing (i.e. health care worker, food service worker);
* Currently suffering from respiratory allergies or a history of seasonal respiratory allergies that are normally active during the study period;
* History of dermatologic disease on the hands, wrists or arms;
* History of 3rd degree burns and/or skin grafts on the hands or wrists;
* History of significant or frequent skin and soft tissue infections;
* Use of androgens, immunomodulators (such as growth factors, systemic corticosteroids, immune globulin, interleukins, interferons) or immunosuppressive medications within 30 days prior to study entry.
* Erythema score of 1.0 and/or dryness scores on the hands at enrollment of greater than Grade 0;
* Subject does not experience colds;
* The subjects from TM&R-0062-08-TXC who were discontinued for irritation, experienced test product related skin reactions or were withdrawn from the study or excluded from the per-protocol analysis for non-compliance.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of rhinovirus-induced common colds. | 9 weeks

SECONDARY OUTCOMES:
Reduction of rhinovirus infections and reduction of common colds. | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Turner, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Jefferson T, Del Mar CB, Dooley L, Ferroni E, Al-Ansary LA, Bawazeer GA, van Driel ML, Jones MA, Thorning S, Beller EM, Clark J, Hoffmann TC, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2020 Nov 20;11(11):CD006207. doi: 10.1002/14651858.CD006207.pub5. PMID 33215698
- [Derived] Turner RB, Fuls JL, Rodgers ND, Goldfarb HB, Lockhart LK, Aust LB. A randomized trial of the efficacy of hand disinfection for prevention of rhinovirus infection. Clin Infect Dis. 2012 May;54(10):1422-6. doi: 10.1093/cid/cis201. Epub 2012 Mar 12. PMID 22412063